CLINICAL TRIAL: NCT00975819
Title: A Phase 2 Study - Clinical Trial Assessing Efficacy and Safety of the mTOR Inhibitor Sirolimus in the Treatment of Complicated Vascular Anomalies
Brief Title: Safety and Efficacy Study of Sirolimus in Complicated Vascular Anomalies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denise Martin Adams (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Denise Martin Adams, Denise Adams, MD/Medical Director, Hemangioma Vascular Malformation Center, Cincinnati Children's Hospital Medical Center, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIR-DA-0901; 5R01FD003712-04 (FDA)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Kaposiform Hemangioendotheliomas; Tufted Angioma; Capillary Venous Lymphatic Malformation; Venous Lymphatic Malformation; Microcystic Lymphatic Malformation; Mucocutaneous Lymphangiomatosis and Thrombocytopenia; Capillary Lymphatic Arterial Venous Malformations; PTEN Overgrowth Syndrome With Vascular Anomaly; Lymphangiectasia Syndromes
MeSH Terms: conditions — Tufted angioma; Lymphangioma; Thrombocytopenia | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Single arm using Sirolimus 0.8 mg/m2 per dose twice daily, Liquid form (1mg/ml) Length: 12 cycles of 28 day cycles
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — liquid dosing based on trough levels
  Other Names: Rapamune; rapamycin

SUMMARY:
The purpose of this study is to determine if the use of sirolimus in the treatment of children and young adults with complicated vascular anomalies will prove to be safe and provide objective response resulting in improved clinical status and quality of life.

Funding Source - FDA OOPD (Food and Drug Administration - Office of Orphan Products Development)

DETAILED DESCRIPTION:
Patients with vascular anomalies (VA) have a spectrum of diseases that can be broadly classified into vascular tumors and malformations. Complicated vascular anomalies can cause disfigurement, chronic pain, and organ dysfunction with significant morbidity and mortality. Despite the severity of potential complications, we lack uniform guidelines for the treatment and response to treatment of children and young adults with these diseases. There are pre-clinical and clinical data supporting the essential regulatory function of the PI3K/Akt/mTOR pathway in vascular growth and organization, and suggest a therapeutic target for patients with complicated vascular anomalies. The overall goal of this trial is to objectively determine the effectiveness and safety of the mTOR inhibitor Rapamycin* in the treatment of children and young adults diagnosed with complicated vascular anomalies. We propose a Phase 2 trial with the diagnostic, therapeutic and response criteria experimentally determined in this study used as a framework for future Phase 3 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Inclusion will be strictly limited to children and young adults with vascular anomalies with complications that require systemic therapy for control.

Diagnosis: All patients must have one of the following vascular anomalies as determined by clinical, radiographic and histologic criteria (when possible):

* Kaposiform Hemangioendotheliomas with Kasabach-Merritt Phenomenon
* Kaposiform Hemangioendotheliomas without Kasabach-Merritt Phenomenon
* Tufted Angioma with Kasabach-Merritt Phenomenon
* Tufted Angioma without Kasabach-Merritt Phenomenon
* Capillary Lymphatico-Venous Malformation (CLVM)
* Venous Lymphatic Malformation (VLM)
* Microcystic Lymphatic Malformation (MLM)
* Multifocal Lymphangiomatosis and Thrombocytopenia (MLT)/Cutaneovisceral Angiomatosis and Thrombocytopenia (CAT)
* Capillary Lymphatic Arterial Venous Malformations (CLAVM)
* PTEN Overgrowth syndrome with vascular anomaly
* Lymphangiectasia Syndromes

If archived tissue is available, histological diagnosis will be confirmed by the pathology lab at the enrolling site.

Complications: Patients must have vascular anomalies that have potential to cause significant morbidity. In addition to the above diagnosis, one or more of the following criteria needs to be met:

* Coagulopathy
* Chronic pain
* Recurrent cellulitis (>3 episodes/year)
* Ulceration
* Visceral and/or bone involvement
* Cardiac dysfunction

Age: Patients must be 0 - 31 years of age at the time of study entry. Enrollment includes patients of both genders and all ethnic groups.

Organ function requirements:

Adequate liver function defined as:

* Total bilirubin (sum of conjugated and unconjugated) ≤1.5 x ULN for age, and
* SGPT (ALT) <5 x ULN for age, and
* Serum albumin > or = 2 g/dL.

Fasting LDL and cholesterol:

* Fasting LDL cholesterol of <160 mg/dL
* Patients taking a cholesterol lowering agent must be on a single medication and on a stable dose for at least 4 weeks

Adequate Bone Marrow Function defined as:

* Peripheral absolute neutrophil count (ANC) > or = 1000/microL
* Hemoglobin > or = 8.0 gm/dL (may receive RBC transfusions)
* Platelet count > or = 50,000/microL (transfusion independent defined as not receiving a platelet transfusion within a 7 day period prior to enrollment)

Note: There is NO platelet requirement for patients with Kasabach-Merritt Phenomenon

Adequate Renal Function Defined as:

• A serum creatinine based on age as follows:

* ≤ 5 years of age maximum serum creatinine (mg/dL) of 0.8
* 6 < age ≤ 10 years of age maximum serum creatinine (mg/dL) of 1.0
* 11 < age ≤ 15 years of age maximum serum creatinine (mg/dL) of 1.2
* > 15 years of age maximum serum creatinine (mg/dL) of 1.5

AND cystatin C equal to or less than the upper limit of normal for the patient. If cystatin C does not initially meet this criterion, it may be repeated or a more sensitive screening by nuclear GFR must be ≥ 70 ml/min.

• Urine protein to creatinine ratio (UPC) < 0.3 g/l

Performance Status: Karnofsky > or = 50 (>10 years of age) and Lansky > or = 50 for patients < or = 10 years of age

Prior therapy requirements:

1. Patients who have undergone surgical resection or interventional radiology procedures for disease control are eligible if they meet all inclusion criteria after surgery/procedure
2. Surgery: At least 2 weeks since undergoing any major surgery
3. Steroids: Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary. Other patients, such as vascular tumor patients, need to be on a weaning dose of steroids (steroid use defined as intravenous or oral steroids required for more than one day).
4. Myelosuppressive chemotherapy: Must not have received within 4 weeks of entry onto this study.
5. Hematopoietic GFs: At least 7 days since the completion of therapy with a GF that supports platelet, red or white cell number or function.
6. Biologic (anti-neoplastic agent): At least 14 days since the completion of therapy with a biologic agent. For agents that have known AEs occurring beyond 14 days after administration, this period must be extended beyond the time during which AEs are known to occur. These patients must be discussed with the Study Chair on a case-by-case basis.
7. Patients diagnosed with Kaposiform Hemangioendotheliomas or Tufted Angiomas will not require a washout period prior to enrollment, but will be required to discontinue the use of prohibited concomitant medications upon enrollment in the study following the guidelines of the protocol.
8. Investigational Drugs: Patients must not have received any non-FDA approved drug within 4 weeks.
9. XRT: > or = 6 months from involved field radiation to vascular tumor.
10. CYP3A4 inhibitors: Patients may not be currently receiving strong inhibitors of CYP3A4, and may not have received these medications within 1 week of entry. (See Appendix II). These include:

    * Macrolide Antibiotics: clarithromycin, telithromycin, erythromycin, troleandomycin.
    * Gastrointestinal prokinetic agents: cisapride, metoclopramide.
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole, clotrimazole
    * Calcium channel blockers: verapamil, diltiazem, nicardipine
    * Other drugs: rifampin, bromocriptine, cimetidine (Tagamet®), danazol, cyclosporine oral solution, lansoprazole (Prevacid®).
    * Grapefruit juice.
11. CYP3A4 inducers: Patients must also avoid strong inducers of CYP3A4, and may not have received these medications within 1 week of entry. These include:

    * Anticonvulsants: carbamazepine, phenobarbital, phenytoin
    * Antibiotics: rifabutin, rifapentine.
    * Herbal preparations: St. John's Wort (Hypericum perforatum, hypericine).
12. Enzyme inducing anticonvulsants: Patients may not be taking enzyme-inducing anticonvulsants, and may not have received these medications within 1 week of entry, as these patients may experience different drug disposition. These medications include:

    * Carbamazepine (Tegretol®)
    * Felbamate (Felbtol®)
    * Phenobarbitol
    * Phenytoin (Dilantinl®)
    * Primidone (Mysoline®)
    * Oxcarbazepine (Trileptal®)

Exclusion Criteria:

* Dental braces or prosthesis only if it interferes with radiologic analysis of vascular anomaly.
* Concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* Chronic treatment with systemic steroids or another immunosuppressive agent. Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary. Patients with the diagnosis of a vascular tumor (KHE, TA) can be on a weaning dose of steroids.
* Patients who require medications that inhibit/induce CYP3A4 enzyme activity to control concurrent medical conditions.
* Known history of HIV seropositivity or known immunodeficiency. Testing is not required unless a condition is suspected.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sirolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A gastric tube or nasogastric tube is allowed.
* Women who are pregnant or breast feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the period they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Women of childbearing potential will be given a pregnancy test within 7 days prior to administration of sirolimus and must have a negative urine or serum pregnancy test.
* Patients who have received prior treatment with an mTOR inhibitor.
* Patients unwilling or unable to comply with the protocol, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Patients who currently have an uncontrolled infection, defined as receiving intravenous antibiotics.

Max Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Adams, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Ricci KW, Hammill AM, Mobberley-Schuman P, Nelson SC, Blatt J, Bender JLG, McCuaig CC, Synakiewicz A, Frieden IJ, Adams DM. Efficacy of systemic sirolimus in the treatment of generalized lymphatic anomaly and Gorham-Stout disease. Pediatr Blood Cancer. 2019 May;66(5):e27614. doi: 10.1002/pbc.27614. Epub 2019 Jan 22. PMID 30672136
- See also: National Organization of Vascular Anomalies — http://www.novanews.org/
- See also: Lymphangiomatosis & Gorham's Disease Alliance — http://www.lgdalliance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened October 2009, closed to enrollment March 2014.
Period: Overall Study
Arm/Group | Sirolimus
Started | 61
Completed | 46
Not Completed | 15
Not completed — Lack of Efficacy | 8
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 8.1 [0.17 to 28.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Overall Response by Radiologic Evaluation, Quality of Life Assessment, and Functional Impairment Score
Description: Measures were determined by 3 distinct methods: radiologic evaluation, functional impairment score (clinical measurement of disease), and health-related quality of life. (HRQOL). The most common radiologic evaluation was MRI but other studies including CT and X-rays were included. HRQOL was assessed using the Pediatric Quality of Life Inventory 4.0 (3-18 years) ad infant Scales (< or = to 2 years) and the Functional Assessment of Chronic Illness System (> 18 years). Third method was the functional impairment score which was adopted from the measure of organ function that have been validated in the quantification of adverse even results from medical therapies and procedures. Patients needed to have complete response, normalization in quality of life and functional impairment score to have a complete response. In order to have a partial response they needed to have improvement in all three areas of assessment and not worsening of any others.
Time Frame: 6 months
Population: Sixty-one patients were enrolled; 57 patients were evaluable for efficacy at the end of course 6.
Measure: Count of Participants; unit: Participants
Groups:
- Sirolimus: Responsiveness to sirolimus by the end of course 6
Arm/Group | Sirolimus
Number analyzed (Participants) | 57
Participants
  Partial Response | 47
  Progressive Disease | 7
  Stable Disease | 3

2. Primary Outcome: Overall Response by Radiologic Evaluation, Quality of Life Assessment, and Functional Impairment Score
Description: as for outcome 1
Time Frame: 12 months
Population: 53 were evaluable at the end of course 12.
Measure: Count of Participants; unit: Participants
Groups:
- Sirolimus: Responsiveness to sirolimus by the end of course 12
Arm/Group | Sirolimus
Number analyzed (Participants) | 53
Participants
  Partial Response | 45
  Progressive Disease | 8

ADVERSE EVENTS:
Groups:
- All Grade 2 and Higher Adverse Events Attributable to Sirolimus: All Grade 2 and Higher Adverse Events Attributable to Sirolimus Per CTCAE Version 3.0, by category
Arm/Group | All Grade 2 and Higher Adverse Events Attributable to Sirolimus
Serious Adverse Events (participants affected / at risk) | 24/61
Other Adverse Events (participants affected / at risk) | 5/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Grade 2 and Higher Adverse Events Attributable to Sirolimus (N=61)
Pain- Abdomen- NOS (General disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Appendix (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 8 (14)
Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Infection- Colon (Infections and infestations) | 1 (1)
CVC port infection (Infections and infestations) | 2 (2)
Airway/ lung (Infections and infestations) | 3 (4)
Immunodeficency (Infections and infestations) | 1 (1)
Phlebitis (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 5 (8)
Weight Loss (General disorders) | 1 (2)
Dehydration (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Grade 2 and Higher Adverse Events Attributable to Sirolimus (N=61)
Blood Bone Marrow (Blood and lymphatic system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No